CLINICAL TRIAL: NCT03640572
Title: Prognostic Value of Disseminated Tumour Cells in Bone Marrow in Patients With Left-sided Colorectal Cancer.
Brief Title: Disseminated Tumour Cells (DTC) in Left Sided Colorectal Cancer (LSCC).
Status: Completed | Type: Observational
Sponsor: Jagiellonian University (Other)
Responsible Party: Principal Investigator, Radoslaw Pach, MD, Ph D, Assisstant Professor, Jagiellonian University
Other Study IDs: DCT LSCC
Record Dates: First submitted 2018-08-17; First posted 2018-08-21 (Actual); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Colorectal Cancer; Bone Marrow Tumor Cell Infiltration
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone Marrow biopsy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Bone Marrow DTC: Patients with left-sided colorectal cancer and disseminated tumour cells in the bone marrow
  Interventions: Diagnostic Test: Bone marrow analysis to identify disseminated tumour cells
- No bone marrow DTC: Patients with left-sided colorectal cancer and no disseminated tumour cells in the bone marrow
  Interventions: Diagnostic Test: Bone marrow analysis to identify disseminated tumour cells

INTERVENTIONS:
Diagnostic Test: Bone marrow analysis to identify disseminated tumour cells — Pelleted cells from bone marrow samples were incubated with an excessive amount of lysing solution for 10 min, repeated 3-4 times to remove erythrocytes. The slides were dried, fixed with a mixture of ethanol and acetone (1 : 1 v v-1), and then stained for 30 min with A45-B/B3 monoclonal antibodies (5 μg ml-1) (Micromet GmbH, Germany), which recognise common epitopes of cytokeratins (CK) including CK 8, 18 and 19.

SUMMARY:
Two metaanalyses of studies on the prognostic significance of circulating cancer cells in colorectal cancer indicated, that the presence of circulating tumour cells (CTC) in the peripheral blood is the negative prognostic factor. However there is no sufficient evidence that disseminated tumour cells (DTC) in the bone marrow of the colorectal cancer patients influence the prognosis. There is the evidence that right-sided and left- sided cancers may have different biology and different prognosis. Therefore in this study the investigators concentrated on the left colon and rectum locations with the locally advanced cancer being the main area of interest.

The aim of this study was to analyse the relation of DTC with the tumor characteristics, cancer progression and survival in left sided colorectal cancer.

DETAILED DESCRIPTION:
A group of 91 colorectal patients treated in a single institution was involved into the study. Only the patients with tumors located in the rectum or left side colon were included. The term left colon was defined as the left 1/3 of transverse colon and all the colon parts distally from this point. None of the colon cancer patients received preoperative chemotherapy, while 5 of the rectal cancer patients received preoperative radiotherapy and two preoperative radiochemotherapy. There were 42 women and 49 men, the mean age 64,7 (SD - standard deviation 10,2). The bone marrow biopsy was performed on the day of surgery after the induction of general anesthesia from posterior superior iliac spine. The 5ml sample of the bone marrow was collected to plastic tubes containing EthyleneDiamineTetraacetic (EDTA). Patients received postoperative chemotherapy if indicated, regardless of their DTC status. All the patients were followed up at least for 5 years or until death.

The incidence of DTC was not related to the depth of infiltration (T feature) being similar in T1-2 and T4 patients. There was no statistically significant difference between the incidence of DTC in N- and N+ patients. The 5 years survival rate for the DTC patients was 59,5% while for the DTC negative patients was 53%.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* histologically proven left-sided colorectal cancer
* signed informed consent

Exclusion Criteria:

* synchronous right sided colon cancer
* history of other neoplasm
* inability to understand and sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with left-sided colorectal cancer operated on in one tertiary centre.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2007-06-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2018-12-30 (Actual)

PRIMARY OUTCOMES:
Overall survival (OS) | 5 years
  OS in patients with and without DTC in bone marrow

SECONDARY OUTCOMES:
Local recurrence rate | 5 years
  Local recurrence in patients with and without DTC in bone marrow
Systemic recurrence | 5 years
  Systemic recurrence in patients with and without DTC in bone marrow

CONTACTS AND LOCATIONS:
Overall Officials: Antoni Szczapanik, Assoc. Prof., Study Chair — Jagiellonian diversity
Locations (1):
- 1st Department of General Surgery, Krakow, Malopolska, Poland